CLINICAL TRIAL: NCT03145363
Title: Mobile Phone Intervention to Reduce Youth Suicide in Rural Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Anthony Pisani, Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: K23MH101449 (NIH)
Record Dates: First submitted 2017-04-25; First posted 2017-05-09 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Help-Seeking Behavior; Emotions; Trusted Adults; Suicide; Positive Affect
MeSH Terms: conditions — Help-Seeking Behavior; Suicide | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Intervention group (receives interactive text messages) and control group (receives informative text messages)
Who Masked: Participant
Masking Description: Participants do not know which group they were randomized into.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): receive interactive text messages
  Interventions: Behavioral: Intervention
- Control (Active Comparator): Receive informational text messages
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Intervention — The intervention group will receive 2-5 interactive text message sequences per week. These messages will invite students to reply using keywords and short free text replies. Messages come from a library of strength-based peer quotations (reviewed for safety), psychoeducational interactions, and games designed to promote emotional skills and use of resources.
  Arms: Intervention
Behavioral: Control — The control group will receive 1-2 (non-interactive) text messages per week containing general SoS concepts (e.g., "Remember: more strengths are better when times get tough").
  Arms: Control

SUMMARY:
The goal of this research project is to conduct a pilot RCT of Text4Strength, an interactive automated text messaging extension of Sources of Strength (SoS), a universal school-based suicide prevention program that prepares diverse 'key opinion leaders' to conduct public health messaging and activities with peers to increase school-wide positive coping norms, communication with trusted adults, and seeking help for suicidal peers (Wyman et al., 2010). The investigators previously developed and field tested Text4Strength messages (RSRB#00047481 and 53924 closed) to demonstrate feasibility, safety, student engagement, and student-perceived relevance for a universal texting extension. The investigators will now conduct a pilot randomized controlled trial in one large school in Western New York that has implemented Sources of Strength for the past two years. The school will continue with Sources of Strength in the 2016-17 school, and add this school-wide texting component as part of this research study. Consistent with Leon's guidelines on pilot studies, the primary focus will be to identify areas of promise, success in reaching proximate targets, and the need for additional modifications (Leon, Davis, & Kraemer, 2011). Findings from this study will inform further refinement of the text messaging program and provide preliminary data for a larger efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

* 9th-12th grade students in study school
* must have own cell phone

Exclusion Criteria:

* no cell phone
* not sufficiently English-speaking to complete surveys

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 222 (Actual)
Dates: Start 2016-06-29 (Actual); Primary Completion 2017-05-26 (Actual); Study Completion 2017-05-26 (Actual)

PRIMARY OUTCOMES:
Emotion self-regulation skills | change from baseline to three-month follow-up
  Difficulties with Emotion Regulation Scales (DERS) (Gratz & Roemer, 2004)
Resources for Coping | change from baseline to three-month follow-up
  uptake of Sources of Strength concepts (Wyman et al., 2010)
Help-Seeking norms | change from baseline to three-month follow-up
  Help-seeking from adults at school (Schmeelk-Cone, et al, 2012)

SECONDARY OUTCOMES:
Depression | baseline, immediate follow-up, three-month follow-up
  Mood and Feelings Questionnaire (MFQ: Angold, et al., 1996; Costello & Angold, 1988)
Suicidal Ideation | baseline, immediate follow-up, three-month follow-up
  one question from the MFQ about suicidal ideation in the past two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anthony R Pisani, PhD, Principal Investigator — University of Rochester Medical Center, Psychiatry Dept

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gould MS, Greenberg T, Munfakh JL, Kleinman M, Lubell K. Teenagers' attitudes about seeking help from telephone crisis services (hotlines). Suicide Life Threat Behav. 2006 Dec;36(6):601-13. doi: 10.1521/suli.2006.36.6.601. PMID 17250466
- [Background] Hahn EA, DeWalt DA, Bode RK, Garcia SF, DeVellis RF, Correia H, Cella D; PROMIS Cooperative Group. New English and Spanish social health measures will facilitate evaluating health determinants. Health Psychol. 2014 May;33(5):490-9. doi: 10.1037/hea0000055. Epub 2014 Jan 20. PMID 24447188
- [Background] Neacsiu AD, Rizvi SL, Vitaliano PP, Lynch TR, Linehan MM. The dialectical behavior therapy ways of coping checklist: development and psychometric properties. J Clin Psychol. 2010 Jun;66(6):563-82. doi: 10.1002/jclp.20685. PMID 20455249
- [Background] Pisani AR, Wyman PA, Petrova M, Schmeelk-Cone K, Goldston DB, Xia Y, Gould MS. Emotion regulation difficulties, youth-adult relationships, and suicide attempts among high school students in underserved communities. J Youth Adolesc. 2013 Jun;42(6):807-20. doi: 10.1007/s10964-012-9884-2. Epub 2012 Dec 18. PMID 23666604
- [Background] Schmeelk-Cone K, Pisani AR, Petrova M, Wyman PA. Three scales assessing high school students' attitudes and perceived norms about seeking adult help for distress and suicide concerns. Suicide Life Threat Behav. 2012 Apr;42(2):157-72. doi: 10.1111/j.1943-278X.2011.00079.x. Epub 2012 Feb 10. PMID 22324773
- [Background] Simons, J. S., & Gaher, R. M. (2005). The Distress Tolerance Scale: Development and Validation of a Self-Report Measure. Motivation and Emotion, 29(2), 83-102. doi:10.1007/s11031-005-7955-3
- [Background] Terwee CB, Roorda LD, de Vet HC, Dekker J, Westhovens R, van Leeuwen J, Cella D, Correia H, Arnold B, Perez B, Boers M. Dutch-Flemish translation of 17 item banks from the patient-reported outcomes measurement information system (PROMIS). Qual Life Res. 2014 Aug;23(6):1733-41. doi: 10.1007/s11136-013-0611-6. Epub 2014 Jan 9. PMID 24402179
- [Background] Wyman PA, Brown CH, LoMurray M, Schmeelk-Cone K, Petrova M, Yu Q, Walsh E, Tu X, Wang W. An outcome evaluation of the Sources of Strength suicide prevention program delivered by adolescent peer leaders in high schools. Am J Public Health. 2010 Sep;100(9):1653-61. doi: 10.2105/AJPH.2009.190025. Epub 2010 Jul 15. PMID 20634440
- [Background] Gratz, K. L., & Roemer, L. (2004). Multidimensional assessment of emotion regulation and dysregulation: Development, factor structure, and initial validation of the difficulties in emotion regulation scale. Journal of Psychopathology and Behavioral Assessment, 26(1), 41-54. doi:10.1023/B:JOBA.0000007455.08539.94
- [Background] Angold, A., Costello, E. J., Messer, S., Pickles, A., Winder, F., & Silver, D. (1996). Development of a short questionnaire for use in epidemiological studies of depression in children and adolescents. International Journal of Methods in Psychiatric Research, 5, 237-249.
- [Background] Costello EJ, Angold A. Scales to assess child and adolescent depression: checklists, screens, and nets. J Am Acad Child Adolesc Psychiatry. 1988 Nov;27(6):726-37. doi: 10.1097/00004583-198811000-00011. No abstract available. PMID 3058677
- [Derived] Pisani AR, Wyman PA, Cero I, Kelberman C, Gurditta K, Judd E, Schmeelk-Cone K, Mohr D, Goldston D, Ertefaie A. Text Messaging to Extend School-Based Suicide Prevention: Pilot Randomized Controlled Trial. JMIR Ment Health. 2024 Dec 6;11:e56407. doi: 10.2196/56407. PMID 39642360